CLINICAL TRIAL: NCT06251882
Title: 6-month Efficacy of Ultrasound-guided Injection of 5% Dextrose for Meralgia Paresthesia
Brief Title: Efficacy of Ultrasound-guided Injection of 5% Dextrose for Meralgia Paresthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhu Jiaan, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB019-001(2)
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Meralgia Paresthetica
Keywords: ultrasound; meralgia paresthetica; D5W
MeSH Terms: conditions — Femoral Neuropathy | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D5W group (Experimental): The patients received one session of ultrasound-guided 10ml D5W injection around the lateral femoral cutaneous nerve as it exited the pelvis.
  Interventions: Other: injection

INTERVENTIONS:
Other: injection — 10ml D5W injection for MP patients

SUMMARY:
Meralgia paresthetica (MP) is one of the most common peripheral entrapment neuropathies of the lower limbs. It is characterized by paresthesia, pain, tingling, numbness, hypersensitivity, or other abnormal skin sensations on the anterolateral aspect of the thigh. The condition results from compression of the lateral femoral cutaneous nerve (LFCN) along its course, often occurring as the nerve exits the pelvis.The injection of 5% dextrose (D5W) under ultrasound guidance is a novel treatment method for peripheral nerve entrapment. However, there is limited evidence about the efficacy of this method for patients with MP. The investigators found D5W was more safe and effective than corticosteroids for patients with MP. Thus, this study aimed to evaluate the 6-month efficacy of ultrasound-guided injection of D5W for MP patients.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 80 years;
* those diagnosed with MP based on clinical and physical examination, with symptoms persisting for at least 3 months;
* a high-resolution ultrasound revealing LFCN compression as it exited the pelvis.

Exclusion Criteria:

* MP resulting from trauma, surgery or occupying lesions affecting the LFCN;
* pregnancy;
* concurrent presence of rheumatic immune diseases, hypothyroidism, or diabetes mellitus;
* a known history of allergy to lidocaine or corticosteroids;
* L2/3 lumbar radiculopathy;
* patients who had undergone local injection or surgery for MP within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale(VAS) | baseline as well as 1month, 3 month, 6 months post-injection
  VAS is one of the most common tool to assess pain severity for patients, ranging from 0(no pain) to 10(most possible pain).

SECONDARY OUTCOMES:
cross-sectional area(CSA) of the nerve | baseline as well as 1month, 3 month, 6 months post-injection
  CSA could reflect the compression of the nerve, to some extent

CONTACTS AND LOCATIONS:
Overall Officials: Jiaan Zhu, Dr, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scholz C, Hohenhaus M, Pedro MT, Uerschels AK, Dengler NF. Meralgia Paresthetica: Relevance, Diagnosis, and Treatment. Dtsch Arztebl Int. 2023 Sep 29;120(39):655-661. doi: 10.3238/arztebl.m2023.0170. PMID 37534445
- [Background] Agarwal N, Mistry JB, Khandge PV, Hansberry DR, Goldstein IM. Meralgia Paresthetica After Spine Surgery on the Jackson Table. Clin Spine Surg. 2018 Mar;31(2):53-57. doi: 10.1097/BSD.0000000000000593. PMID 29135610
- [Background] Wu YT, Ke MJ, Ho TY, Li TY, Shen YP, Chen LC. Randomized double-blinded clinical trial of 5% dextrose versus triamcinolone injection for carpal tunnel syndrome patients. Ann Neurol. 2018 Oct;84(4):601-610. doi: 10.1002/ana.25332. Epub 2018 Oct 4. PMID 30187524